CLINICAL TRIAL: NCT06712745
Title: Feasibility Study of Personalized Ultra-fractionated Stereotactic Ablative Radiotherapy (PULSAR) for Cancers of the Central Lung
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Principal Investigator, Kenneth Westover, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-1215
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-05

CONDITIONS: Cancer, Lung; Metastasis
Keywords: lung; central lumg; cancer; metastasis; PULSAR; non small cell lung cancer; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — DEAE-Dextran

STUDY DESIGN:
Intervention Model Description: Study agent:Stereotactic ablative body radiation (SABR)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility (Experimental): Patients treated with PULSAR will undergo treatment over a total duration of 2-5 months with 3-4 weeks between each fraction. PULSAR treatments completed within 6 months will be acceptable if treatment breaks are required. In the event of a complete response between fractions, remaining fractions will be withheld at the discretion of the treating physician. Treatment may also be terminated for selected grade 3 or higher AEs. Treatment may also be terminated for regional or systemic progression detected during the PULSAR treatment interval.
  Interventions: Radiation: Personalized Ultra-fractionated stereotactic ablative radiotherapy (PULSAR)

INTERVENTIONS:
Radiation: Personalized Ultra-fractionated stereotactic ablative radiotherapy (PULSAR) — Radiation Therapy Prescription Dose: A dose of 40-50 Gy in 5 fractions prescribed to the PTV will be used for all cases

SUMMARY:
The objective of this study is to enhance the safety profile of SAbR in ultra-central tumors of the lung (primary or metastatic) without compromising its effectiveness.

DETAILED DESCRIPTION:
This will be achieved by demonstrating the feasibility of applying adaptive radiation therapy given in PULSAR fractionation and using a 1.5T MR-guided linac system with real-time motion monitoring (Unity, Elekta). The hypothesis is that safety can be improved through: (1) better visualization of tumors, leading to less uncertainty when delineating GTVs; (2) reduced margins for setup, motion, or other sources of uncertainty; and (3) improved normal tissue healing between radiation fractions. To achieve this, we propose a personalized ultrafractionated stereotactic adaptive radiotherapy (PULSAR) delivery schedule, administering 5 fractions total, given as one fraction every 3 weeks (Fig. 3) and using MRI-guided adaptive treatment planning.

This study is single arm in nature and in the feasibility phase

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Histologically proven diagnosis of cancer. At a minimum, the lung tumor in consideration for treatment must be clinically judged as related to the biopsied site.
3. Stage: Tumor (ITV) 1.5 - 5 cm in maximum diameter.
4. Tumor entirely within the 2 cm "central zone" or within 1 cm of the mediastinum, esophagus or proximal bronchial tree by investigator assessment.
5. Zubrod/ECOG Performance Status 0-2 within 30 days prior to registration.
6. Ability to tolerate MRI.
7. All men, as well as women of child-bearing potential* must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of consent, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Note: A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
2. Plans for the patient to receive other local therapy in lung (including standard fractionated radiotherapy and/or surgery) while on this study, except at disease progression.
3. Females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry.
4. Prior administration of anti-VEGF (vascular endothelial growth factor) therapy within 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy- Survivability and response | 4 years
  Rates of overall response will be assessed by RECIST criteria.Efficacy will be compared between PULSAR and historical controls from HILUS using ANOVA and chi-square test.
  Kaplan-Meier methods will be used to estimate progression-free survival, time to subsequent SABR, overall survival, clinical benefit rate, time to treatment discontinuation, duration of response, and time to new metastases.
  Response duration will be summarized for patients who responded. Descriptive summary statistics such as median and interquartile range (25% and 75% percentiles) will be used.

SECONDARY OUTCOMES:
Change in Tumor Volume | 1 year
  Change in tumor volume will be measured by comparing pre-treatment tumor volume to during-treatment tumor volumes as measured by MRI and will be analyzed using an independent t-test.

OTHER OUTCOMES:
Dosimetry | 1 year
  Dosimetry will be compared for relevant OARs, including heart, esophagus, and lung, and will be analyzed using an independent t-test.

CONTACTS AND LOCATIONS:
Overall Officials: KENNETH WESTOVER, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States